CLINICAL TRIAL: NCT07057232
Title: Estimating the Prevalence of Chronic Insomnia in Patients With Non-cancer Chronic Pain
Brief Title: Chronic Insomnia in Non-Cancer Pain Patients
Acronym: PainSomnia
Status: Recruiting | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Societat Catalana de Dolor (Catalan Society for Pain) (Unknown); Hospital del Mar (Other)
Responsible Party: Sponsor
Other Study IDs: SCD-2024-01
Record Dates: First submitted 2025-06-27; First posted 2025-07-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Non-cancer Pain; Insomnia
Keywords: Insomnia; Chronic non-cancer pain; Prevalence
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic non-cancer pain patients: Adult non-cancer chronic pain patients receiving care in outpatient settings from a pain specialist or within a dedicated pain unit.
  Interventions: Other: Usual care provided from pain specialist or within a dedicated pain unit

INTERVENTIONS:
Other: Usual care provided from pain specialist or within a dedicated pain unit — Adult non-cancer chronic pain patients receiving care in outpatient settings from a pain specialist or within a dedicated pain unit
  Other Names: Standard care

SUMMARY:
Pain and sleep are closely linked physiological processes that support overall health and functioning. Increasing evidence shows a dynamic, bidirectional relationship: poor sleep increases pain sensitivity, while chronic pain disrupts normal sleep. Both conditions are highly prevalent and significantly impair quality of life, making them major public health concerns.

Chronic pain, defined as pain lasting more than three months, affects around 17% of adults in Spain. Insomnia, though common, is harder to define due to its overlap with medical and psychiatric conditions. It may present as a symptom, a syndrome, or a formal sleep disorder, leading to variability in prevalence estimates.

Current diagnostic criteria, including DSM-5 and the International Classification of Sleep Disorders, Third Edition (ICSD-3), adopt the unified concept of chronic insomnia disorder, defined as persistent difficulty with sleep initiation, maintenance, or quality, despite adequate opportunity for sleep, and associated with daytime impairment.

ICSD-3 distinguishes three types of insomnia:

* Chronic insomnia disorder: symptoms ≥3 times/week for ≥3 months;
* Short-term insomnia disorder: symptoms lasting less than 3 months;
* Other insomnia disorder: symptoms not meeting criteria for the above.

About one-third of the general population reports insomnia symptoms. However, when both night symptoms and daytime impact are considered, the prevalence of chronic insomnia disorder is estimated at 6-10%. Women are more frequently affected, with a female-to-male ratio of about 1.4:1.

Despite this, few studies have assessed insomnia specifically in people with chronic non-cancer pain. This gap is important, as untreated insomnia may worsen pain and reduce treatment efficacy, reinforcing a vicious cycle.

This observational study (PainSomnia) aims to estimate the prevalence of chronic insomnia among adults with chronic non-cancer pain. The results will help support integrated, individualized treatment approaches that address both sleep and pain in this high-risk population.

DETAILED DESCRIPTION:
Sleep and pain are two biologically and evolutionarily significant processes that play a fundamental role in maintaining health and protecting bodily function. These processes interact through a delicate physiological balance. Although the exact mechanisms underlying the relationship between pain and sleep are still under investigation, current evidence supports a dynamic and bidirectional interaction between the two. Pain can disrupt sleep and reduce its capacity to provide necessary physiological and mental recovery. Conversely, inadequate or fragmented sleep can worsen existing pain conditions or contribute to the development of new pain syndromes, further impairing sleep continuity and quality.

Due to their high prevalence and impact on health and daily functioning, chronic pain and insomnia represent two major public health challenges and are associated with substantial economic and social costs.

Chronic Pain Chronic pain is typically defined as pain that persists for longer than three months and is associated with significant emotional distress, functional impairment, or both. The Pain Proposal, a European initiative aimed at understanding the burden of chronic pain, estimated that approximately 19% of the European population is affected by chronic pain. In Spain, the estimated prevalence is slightly lower, at around 17%. The economic burden of chronic pain is considerable-estimated at over €300 billion annually across Europe, accounting for roughly 1.5% to 3% of GDP. In Spain, the national cost is estimated at €16 billion annually, or approximately 2.5% of GDP.

Chronic pain has a profound negative impact on patients' quality of life, affecting physical health, emotional well-being, and social, familial, and occupational functioning. Comorbidities are common. In Spain, approximately 47% of patients with chronic pain also experience depression, and 50% report sleep disturbances. Sleep disturbances in this context encompass a range of conditions, including difficulties with sleep initiation and maintenance, as well as abnormal events during sleep such as sleep apnea, restless legs syndrome, and insomnia.

Insomnia The diagnostic criteria for insomnia have undergone significant revisions in recent years. Both the DSM-5 and the ICSD-3 have simplified and unified the diagnostic categories, moving toward a more clinically relevant concept of chronic insomnia disorder.

According to ICSD-3, chronic insomnia is characterized by persistent difficulties in initiating or maintaining sleep, or experiencing restorative sleep, occurring at least three times per week for at least three months, despite adequate sleep opportunity and conditions. These disturbances must cause clinically significant distress or impairment in social, occupational, educational, academic, or other important areas of functioning. The thresholds used to define clinical significance-such as sleep onset latency or wakefulness after sleep onset greater than 20 minutes in youth or 30 minutes in older adults-are generally based on subjective reports and clinical observation.

Chronic Pain and Insomnia: A Bidirectional Relationship Historically, insomnia was viewed as a secondary consequence of chronic pain. However, more recent research highlights a bidirectional relationship, where each condition may contribute to and exacerbate the other. Pain can fragment sleep, while disrupted sleep reduces pain thresholds and can trigger spontaneous pain episodes.

Insomnia may act as both a trigger and a perpetuating factor in chronic pain. A landmark sleep deprivation study conducted in 1999 at the University of Washington found that women subjected to selective sleep deprivation exhibited decreased pain tolerance. Since then, multiple studies have confirmed that individuals with insomnia exhibit heightened sensitivity to experimental pain stimuli.

There is strong evidence that short or disrupted sleep can induce hyperalgesia. Additionally, chronic sleep loss has been shown to predict the onset or worsening of chronic pain conditions. Longitudinal studies further support the idea that sleep problems in individuals without existing pain may significantly increase the risk of developing chronic pain syndromes.

The central nervous system has built-in mechanisms to preserve sleep, including neural filtering at the brainstem and descending inhibitory pathways designed to suppress the arousing effects of incoming sensory information. However, pain can override these mechanisms, disrupting both the continuity and architecture of sleep. The extent of this disruption depends on both the intensity of nociceptive stimuli and the individual's susceptibility to sleep fragmentation.

Clinical Relevance and Research Gap Patients with chronic pain are at significantly higher risk for insomnia compared to individuals without pain. The interaction between chronic pain and chronic insomnia is best understood as a vicious cycle in which each condition amplifies the other.

Current clinical guidelines advocate for a multidisciplinary approach to managing chronic pain, which includes addressing associated conditions such as insomnia. Failing to treat insomnia in this population can create a major barrier to effective pain management.

Despite the high co-occurrence of these conditions, no studies to date have quantified the prevalence of chronic insomnia among patients with chronic non-cancer pain in the Spanish population. Although prior studies have estimated the prevalence of sleep disturbances in chronic pain populations to range from 50% to 90%, these estimates vary widely depending on definitions used and have not been validated in local cohorts.

Understanding the true burden of insomnia in this population is essential for developing targeted therapeutic strategies that can alleviate symptoms and prevent deterioration in quality of life. This study, PainSomnia, is designed to fill this knowledge gap by providing reliable, population-specific data on the prevalence of chronic insomnia in adults with chronic non-cancer pain.

The results of this study are expected to inform the design of integrated care pathways and public health policies, ensuring that comorbid insomnia is identified early and managed appropriately in individuals with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Either biological sex
* Diagnosed with chronic non-cancer pain
* Receiving care in a pain unit or by a pain specialist
* Able to understand and participate in the study
* Who sign informed consent

Exclusion Criteria:

* Deemed unable or unlikely to cooperate adequately with study procedures at the discretion of the pain specialist or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult non-cancer chronic pain patients receiving care in outpatient settings from a pain specialist or within a dedicated pain unit.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with chronic non-cancer pain and insomnia | At a single time point during the baseline visit.
  Chronic insomnia will be assessed based on participants' self-reports. A positive screening will require affirmative responses to all five diagnostic criteria (Criteria A-E) for insomnia disorder, as defined by the ICSD-3 Diagnostic Criteria for Insomnia Disorder, as well as confirmation that sleep initiation or maintenance difficulties occur more than three times per week and have persisted for at least three months.
  For participants reporting chronic insomnia, severity will be evaluated using the Insomnia Severity Index (ISI), a validated 7-item questionnaire with total scores ranging from 0 to 28. The global ISI score is interpreted as follows: 0-7: no clinically significant insomnia; 8-14: subthreshold insomnia; 15-21: clinical insomnia (moderate severity); 22-28: clinical insomnia (severe) (Bastien, 2001).

SECONDARY OUTCOMES:
Proportion of patients with chronic non-cancer pain and moderate/severe pain intensity (>4). | At a single time point during the baseline visit.
  Pain intensity will be assessed using a 0-10 Numerical Rating Scale (NRS), where 0 indicates no pain and 10 represents the worst pain imaginable. Moderate to severe pain is defined as a score greater than 4, based on the patient's reported worst pain during the past week.
Proportion of patients with moderate to severe chronic non-cancer pain intensity, and chronic insomnia. | At a single time point during the baseline visit.
  This outcome combines pain and sleep criteria. Patients must meet both the chronic insomnia criteria (ICSD-3 + ISI) and report a pain score >4 on the NRS to be included.
Proportion of patients with poor sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI) | At a single time point during the baseline visit
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a validated 19-item self-reported questionnaire that assesses sleep disturbances over the past month across seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The global score ranges from 0 to 21. A global score greater than 5 will be used to identify patients with poor sleep quality, based on established sensitivity (89.6%) and specificity (86.5%) thresholds (Buysse et al., 1989).
Proportion of patients with chronic non-cancer pain and clinically significant anxiety | At a single time point during the baseline visit
  Anxiety will be assessed using the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS), a validated 14-item self-administered questionnaire. Seven items measure anxiety, with scores ranging from 0 to 21. A score of 11 or higher indicates clinically significant anxiety.
Proportion of patients with chronic non-cancer pain, chronic insomnia, and clinically significant anxiety | At a single time point during the baseline visit
  This outcome identifies the proportion of patients who meet diagnostic criteria for both chronic insomnia (based on ICSD-3 criteria and ISI score) and clinically significant anxiety (HADS anxiety subscale score ≥11).
Proportion of patients with chronic non-cancer pain and clinically significant depression. | At a single time point during the baseline visit.
  Depression will be assessed using the depression subscale of the Hospital Anxiety and Depression Scale (HADS). Seven items measure depressive symptoms.
Proportion of patients with chronic non-cancer pain and positive mood. | At a single time point during the baseline visit.
  Mood will be assessed using the Spanish version of the Profile of Mood States (POMS), a 44-item self-reported questionnaire that evaluates six conceptual mood dimensions: Anger (11 items), Fatigue (6), Vigor (5), Friendship (6), Tension (7), and Depressed Mood (9). Each item is scored on a 5-point Likert scale from 0 ("not at all") to 4 ("extremely"). Positive mood will be operationalized based on higher scores in the Vigor and Friendship subscales.
Proportion of patients with chronic non-cancer pain, chronic insomnia, and clinically significant depression. | At a single time point during the baseline visit.
  This outcome identifies the proportion of patients who meet criteria for both chronic insomnia (per ICSD-3 and ISI) and clinically significant depression (HADS depression subscale score ≥11).
Proportion of patients with chronic non-cancer pain, chronic insomnia, and positive mood. | At a single time point during the baseline visit.
  This outcome refers to the proportion of patients with both chronic non-cancer pain and chronic insomnia (per ICSD-3 criteria and ISI) who also demonstrate a positive mood, as measured by the Vigor and Friendship subscales of the POMS questionnaire (Spanish version) (Andrade, 2010). Positive mood is defined by higher scores on these subscales, rated on a 0-4 Likert scale.
Proportion of patients with chronic non-cancer pain and reduced well-being or functional capacity. | At a single time point during the baseline visit.
  Health-related quality of life will be assessed using two validated instruments. The SF-12 measures physical and mental health across eight domains using 12 items derived from the SF-36. Scores reflect well-being and functional status. The EQ-5D-3L evaluates five health dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each with three severity levels. Patients reporting moderate or severe problems in at least one EQ-5D-3L domain or scoring low on SF-12 will be classified as having reduced well-being or functional capacity.
Proportion of patients with chronic non-cancer pain, chronic insomnia, and reduced well-being or functional capacity. | At a single time point during the baseline visit.
  Among patients with chronic pain and chronic insomnia (per ICSD-3 and ISI), quality of life will be evaluated using the SF-12 and EQ-5D-3L. The SF-12 includes 12 items across eight health dimensions, and the EQ-5D-3L assesses five domains with three levels of severity. Patients reporting moderate or severe impairment in any EQ-5D-3L domain or low SF-12 scores will be categorized as having reduced well-being or functional capacity.
Proportion of patients with chronic non-cancer pain who use benzodiazepines or hypnotic medications. | At a single time point during the baseline visit.
  This outcome captures the proportion of participants with chronic non-cancer pain who report current use of benzodiazepines and/or hypnotic medications at the time of assessment. Medication use will be self-reported by the participant during the baseline visit. Results will be presented as number and percentage of users.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Montes Pérez, MD, PhD, Principal Investigator — Hospital del Mar
Locations (15):
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Instituto de Medicina y Cirugía, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Catalonia
  - Hospital de Viladecans, Hospitalet Del Llobregat, Catalonia
  - Hospital Universitari de Bellvitge, Hospitalet Del Llobregat, Catalonia
  - Centre Avantmèdic Ponent, Lleida, Catalonia
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia
  - Complex Hospitalari Moisés Broggi, Sant Joan Despí, Catalonia
  - Hospital Universitari Joan XXIII, Tarragona, Catalonia
  - Hospital Universitari Sant Joan de Reus, Tarragona, Catalonia
  - Hospital de Tortosa Verge de la Cinta, Tarragona, Catalonia
  - Consorci Sanitari de Terrassa, Terrassa, Catalonia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available by the principal investigator upon reasonable request and subject to approval, in accordance with applicable data protection and ethical guidelines.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be made available 6 months after study completion and will remain available for up to 5 years upon request.
Access Criteria: Qualified researchers may request access to de-identified IPD for secondary analyses that are consistent with the original study objectives. Requests must include a research proposal and data use agreement, and will be reviewed by the principal investigator. Data will be shared in compliance with applicable ethical and legal standards.

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246